CLINICAL TRIAL: NCT00175734
Title: Integrated Studies in Vascular Reactivity and Anemia Correction Therapy in Endstage Kidney Disease Patients
Brief Title: Interactive Studies of Endstage Diabetic Dialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04-0007
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes
Keywords: Vascular Reactivity; Anemia Correction Therapy; Hemodialysis patients; Diabetic and non-diabetic patients; Diabetes in Hemodialysis patients
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: High Hemoglobin Concentration — The purpose of this study is to document relevant and related clinical changes associated with different hemoglobin concentrations in diabetic hemodialysis patients.
Procedure: Low Hemoglobin Concentration — The purpose of this study is to document relevant and related clinical changes associated with different hemoglobin concentrations in diabetic hemodialysis patients.

SUMMARY:
The purpose of this study is to document relevant and related clinical changes associated with different hemoglobin concentrations in diabetic hemodialysis patients.

Hypothesis: The expansile capacity of blood vessels is affected by different hemoglobin concentrations in diabetic hemodialysis patients.

DETAILED DESCRIPTION:
Vascular disease is an important cause of morbidity and mortality in patients with chronic kidney disease (CKD), of which a large proportion is diabetic. Diabetics have complex and multiple reasons for vascular disease, and there is accumulating evidence of associated poor endothelial cell function, particularly in those with kidney disease. One important mechanism through which this might occur relates to changes in shear rate and stress resulting from different viscosity levels. Such fluctuations are increasingly recognized to affect endothelial cell function and hence vessel-wall adaptability in both the short and long term.

Little is known of the consequence of different shear effects on endothelial cell function at various hemoglobin levels in kidney disease. There is some evidence to suggest however that, in the presence of micro-vascular disease, a relative anemia, with associated lower viscosity and shear stress, may be of benefit compared to higher hemoglobin levels.

Diabetics account for almost 40% of dialysis patients worldwide, and are the fastest growing component of the epidemic of CKD. Thus, an understanding of optimal treatment targets for anemia therapy, and the impact of different target levels of hemoglobin on vascular wall function is imperative.

ELIGIBILITY:
Inclusion Criteria:

* Diabetics and non-diabetics on hemodialysis
* On erythropoietin and iron
* On a statin

Exclusion Criteria:

* Uncontrolled blood pressure (BP)
* Ulcers
* Amputations
* Unstable cardiac function
* Malignancy
* Planned operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To determine what hemoglobin level is best for diabetic dialysis patients. Specific parameters: endothelial cell function and related expansile capacity of blood vessels. *Assessed through labs and pulse wave velocity test | 8-12 months per participant

SECONDARY OUTCOMES:
Pulse rate, BP, respiratory rate, peripheral oxygen saturation, ECG during 6-min walk-test and Health Related Quality of Life Assessment as measured by questionnaires | 8-12 months per participant

CONTACTS AND LOCATIONS:
Overall Officials: Adeera Levin, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada